CLINICAL TRIAL: NCT03252626
Title: Study on the Efficacy of Alprostadil Injection in Patients With Acute Ischemic Stroke
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SEAAIS
Record Dates: First submitted 2017-08-08; First posted 2017-08-17 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-02

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Alprostadil; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alprostadil (Active Comparator): Based on the standard medical care, 2ml of Alprostadil
  Interventions: Drug: Alprostadil
- Normal saline (Placebo Comparator): Based on the standard medical care, 2ml of 0.9% saline as the placebo
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Alprostadil — Alprostadil injection USP for intravascular infusion contains 500 micrograms Alprostadil, more commonly known as prostaglandin E1. Vasodilation, inhibition of platelet aggregation are among the most notable of these effects.
  2ml Alprostadil injection added into 10ml 0.9% saline.
  Arms: Alprostadil
Drug: Normal saline — 2ml normal saline injection added into 10ml 0.9% saline.
  Arms: Normal saline

SUMMARY:
Ischemic stroke has a variety of treatments and currently drug therapy is one of the main treatments.A number of clinical studies have proved that alprostadil (PGE1) has pharmacological effects of significant dilation of blood vessels, inhibition of plate aggregation, anti-atherosclerosis and increased cerebral blood flow.Evaluate the 90-days efficacy by comparing two groups of patients'(one with alprostadil,another with placebo) mRS.

ELIGIBILITY:
Inclusion Criteria:

1. ischemic stroke diagnosed by CT or MRI
2. Age: 18-75 years
3. Pre-stroke mRS score is 0-1
4. within 72 hours symptoms onset
5. 4 ≤ NIHSS <20
6. Patient is willing to participate voluntarily and to sign a written patient informed consent

Exclusion Criteria:

1. intracranial tumors, encephalitis or lesions diagnosed by CT or MRI
2. patients with thrombolytic therapy
3. low platelet , blood system diseases or other bleeding tendency
4. suspected subarachnoid hemorrhage or aortic dissection coma
5. atrial fibrillation, myocardial infarction, heart valve disease, infective endocarditis, heart rate <50 beats / min
6. ALT or AST continued to rise more than 3 times the upper limit of normal creatinine clearance rate<30ml/min
7. Dementia and mental illness
8. Patient who is participating in other trials or has been participated in other trials in recent 3 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 950 (Estimated)
Dates: Start 2024-04-18 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale at Day 90 | day 90

SECONDARY OUTCOMES:
Incidence of major vascular events in 30 or 90 days including ischemic stroke and hemorrhagic stroke | day 30, day 90
  Major adverse vascular events include ischemic stroke, hemorrhagic stroke, TIA, myocardial infarction and vascular-related death.
Incidence of stroke events in 30 or 90 days including ischemic stroke and hemorrhagic stroke | day 30, day 90
Barthel Index score | day 30, day 90
  compared the changes in activities of daily living (Barthel index) between the two groups
EQ-5D scale | day 30, day 90
  compared the changes in EQ-5D scale
Documentation of adverse events (AEs) | day 30, day 90
  compared the rates of adverse events